CLINICAL TRIAL: NCT02612441
Title: The Efficacy of Acupuncture on Patients With First Acute Ischemic Stroke, With Signs of Hemiplegia and Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acupuncture_neurology_CTIL
Record Dates: First submitted 2015-11-10; First posted 2015-11-23 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 real Acupuncture group-intervention (Experimental): real Acupuncture Needles
  Interventions: Device: real Acupuncture Needles
- 2 sham Acupuncture group (Sham Comparator): sham Acupuncture Needles
  Interventions: Device: sham Acupuncture Needles

INTERVENTIONS:
Device: real Acupuncture Needles — Acupuncture needles
  Arms: 1 real Acupuncture group-intervention
Device: sham Acupuncture Needles — sham Acupuncture Needles
  Arms: 2 sham Acupuncture group

SUMMARY:
Chinese Acupuncture can improve the motor ability of patients after having first acute ischemic stroke, in time scale up to 3 weeks from when the ischemic stroke occur and in minimum receiving number of 3 Acupuncture treatments.

The accepted treatment on cerebral vascular accident (CVA) is focus on two lines: the first is the treatment when the stroke occurs, and the second is prevention from having more cerebral vascular accident in the future.

In the first accepted treatment line, the only medicinal measure that stand up in critique of organized researches, is Tissue Plasminogen Activator (TPA), and there is Short and limited time after the CVA occur that it can be used. Also (TPA) can be used only on part of the patients with specific defined criterions.

The aim of this study is to add a new accepted treatment method that appointed to improve the results of acute ischemic stroke by Chinese Acupuncture. The written works on this topic is unambiguously.

DETAILED DESCRIPTION:
The number of participant in the clinical trial: approximately 100 patients. 50 patients will receive Chinese Acupuncture and the others 50 will receive sham Acupuncture.

Stages and work method:

The treatments in Acupuncture will occur every week. Each patient will receive minimum 3 Acupuncture/ sham treatments while staying in the neurology department.

1 After the suitable patients selected to be included in the study, with the assistance of statistical software, the acupuncturist will get from each patient approval to be participating in the study.

2. The direct physician of all the patients that will be participate in the study will approve the accepted treatment in Acupuncture/ sham and get the patients acceptance by signature.

3. The acupuncturist will receive a list of all the patients after they signed the research agreement forms, and after they have been taking The National Institutes of Health Stroke Scale- (NIHSS) and Medical Research Council (MRC) Scale for Muscle Strength..

4. The first treatment for each patient from each group (real or sham acupuncture), will take approximately 45 minutes and include:

1. the acupuncturist will filling an intake form, according to the principle of Chinese medicine
2. treatment: Staying with needles / sham needles for about 20 minutes. *take notice that the following treatments will take approximately 30 minutes and includes filling brief questions form according to the principle of Chinese medicine and treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients with first acute ischemic stroke, with preserved cognitive awareness and with the ability to sign on the research agreement forms.

Division for two main groups:

* Group number 1: will get real Acupuncture
* Group number 2: will get false Acupuncture- ( SHAM).

  * The patients will be selected with the assistance of statistical software which will divide them randomly and equally by the standard Criteria.

Exclusion Criteria:

* Patients with understanding dysfunction:

  * Dysphasia, sensory aphasia,
  * Patients with cerebral hemorrhage,
* pregnant women's, children's, and Patients with lack of judgment ability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-10-22 (Actual)

PRIMARY OUTCOMES:
(NIHSS) | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical center, Neurology Department, Haifa, Israel